CLINICAL TRIAL: NCT02810977
Title: Ultrasound Assessment of Gastric Content and Volume After Complete Fasting in Patients Undergoing Surgery at Two University Hospitals: A Multicentric Study
Brief Title: Ultrasound Assessment of Gastric Content and Volume
Status: Completed | Type: Observational
Sponsor: Fundación Santa Fe de Bogota (Other)
Collaborators: Hospital Universitario San Ignacio (Other)
Responsible Party: Principal Investigator, Jose Alejandro Valencia, MD, Fundación Santa Fe de Bogota
Other Study IDs: CCEI-5325-2016
Record Dates: First submitted 2016-06-17; First posted 2016-06-23 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Fasting
Keywords: gastric volume; gastric content; ultrasound; perioperative fasting
MeSH Terms: conditions — Fasting | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Ultrasound — Ultrasound assessment of gastric content and volume

SUMMARY:
Anesthesiologists try to avoid complications with significant peri -operative morbidity and mortality such as bronchoaspiration in patients requiring a surgical procedure under anesthesia. Currently, this is achieved based on experts recommendations from the American Society of Anesthesiologists. However, there are tools like ultrasound that allow assessment of gastric content and volume. This tool allows to individualize each patient and base the decisions objectively. The investigators will assess gastric content and volume by ultrasound in patients who have fasted and require surgery at two University Hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years
* perioperative fasting time between 8 and 14 hours
* American Society of Anesthesiologists status I, II, III
* Scheduled surgery

Exclusion Criteria:

* Abdominal pathology surgical emergency
* Unable to adopt right lateral decubitus position
* Altered gastrointestinal tract anatomy excluding hiatal hernia
* Body mass index greater than 40
* Patients on enteral nutrition probe or with nasogastric probe
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women 18 years or older requiring surgery with complete preoperative fasting (more than 8 hours but less than 14), ASA I-III.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Gastric content | June to December
  Ultrasound assessment of gastric content (empty, fluids, or solid) of patients undergoing surgery after complete fasting (more than 8 hours)
Gastric volume | June to December
  Ultrasound assessment of gastric volume (in milliliters) of patients undergoing surgery after complete fasting (more than 8 hours)

SECONDARY OUTCOMES:
Association of gastric content and volume with special conditions as assessed by Anova or Kruskal as appropriate | June to December
  To identify the association between gastric content and volume with conditions such as diabetes, obesity, hiatal hernia, among others.
Association with fasting time | June to December
  To identify the association between gastric content and volume and preoperative fasting time.

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Valencia, MD, Principal Investigator — Fundacion Santa Fe de Bogota
Locations (2):
- Colombia (2):
  - Hospital Universitario Fundacion SantaFe de Bogota, Bogotá, Bogota D.C.
  - Hospital Universitario San Ignacio, Bogotá, Bogota D.C.

IPD SHARING:
Plan to Share IPD: Yes